CLINICAL TRIAL: NCT00865644
Title: Pilot Study of Topical Imiquimod 5% Cream for Treatment of Cutaneous Neurofibromas in Adults With Neurofibromatosis 1
Brief Title: Topical Imiquimod 5% Cream for Treatment of Cutaneous Neurofibromas in Adults With Neurofibromatosis 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Scott Randall Plotkin, MD, PhD, Associate Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 08-347
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2017-01-10 (Estimated); Status verified 2017-01

CONDITIONS: Neurofibromatosis Type 1; Cutaneous Neurofibromas
Keywords: imiquimod 5% cream
MeSH Terms: conditions — Neurofibromatosis 1 | interventions — Imiquimod

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imiquimod (Experimental)
  Interventions: Drug: Imiquimod 5% Cream

INTERVENTIONS:
Drug: Imiquimod 5% Cream — Applied topically to three tumors 5 times per week for a full 6 weeks

SUMMARY:
The purpose of this study is to determine if imiquimod cream can reverse the growth of neurofibromas. Imiquimod is a skin cream that works by stimulating the body's immune system to respond to tumors. Imiquimod cream is approved for use in patients with various skin lesions, including actinic keratosis, superficial basal cell carcinoma, and external genital warts. Information from these studies, as well as previous laboratory studies, suggest that imiquimod cream may help shrink neurofibromas or keep them from growing.

DETAILED DESCRIPTION:
* Three of the participant's tumors will be treated with imiquimod cream and one tumor (out of all the remaining tumors) will be followed without treatment (control tumor).
* Participants will be given a tube of imiquimod cream and be asked to apply it to the three tumors 5 times per week, for a full 6 weeks (Monday through Friday).
* Participants will be required to come to the hospital for examinations on Week 1, 2, 4 and 6 (+/- 3 calendar days) and after their last dose of imiquimod cream on Weeks 9, 12 and 18 (+/- 5 calendar days. The following tests and procedures will be performed: skin test; vital signs and measurements and photographs of the tumors. Participants will be asked to participate in an optional skin biopsy on Week 4 and research blood tests wil lbe taken on Day 1.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of NF1 based on NIH criterial with two or more of the following characteristics:

  * six or more cafe-au-lait macules (1.5cm or greater in size)
  * skin fold freckling in the axilla or groin
  * optic pathway glioma
  * two or more Lisch nodules of the iris
  * distinctive bony lesions such as dysplasia of the sphenoid wing or of a long bone such as the tibia
  * two or more neurofibromas of any type of 1 or more plexiform neurofibroma
  * first degree relative with NF1
* Participants must have at least four cutaneous neurofibromas on skin exam with the following qualities:

  * the lesion must be discrete by clinical exam and must not be contact with another skin tumor
  * the lesion must be amenable to measurement with calipers with minimum dimension of 5mm and maximum dimension of 30mm
  * the lesions must be located on the trunk, neck, or extremities (excluding the hands and feet) and must be located in an area that can be photographed
  * histologic confirmation of tumor type is not required in the setting of compatible clinical setting
* No treatment with an investigation agent for cutaneous neurofibromas within the last 3 months
* 18 years of age or older

Exclusion Criteria:

* Pregnant and nursing women
* Patients who have had chemotherapy or radiotherapy within 6 weeks prior to entering the study or those who have not recovered from adverse events due to agents administered more than 6 weeks earlier
* Patients may not be receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to imiquimod
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-03; Primary Completion 2010-04 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
To determine the effect of topical imiquimod 5% cream on tumor volume of cutaneous neurofibromas in adult subjects with neurofibromatosis 1 | 2 years

SECONDARY OUTCOMES:
To correlate the inflammatory infiltrate adjacent to treated lesions during treatment with tumor response and to determine the number of circulating Tregs in this patient population | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Scott R. Plotkin, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States